CLINICAL TRIAL: NCT00138268
Title: Pilot Study to Optimize and Standardize Umbilical Cord Blood Collection and the Isolation, Freezing and Transportation of Cells for Studies of Cellular Immune Responses to Immunization
Brief Title: Pilot Study Freeze and Transport Immune Cells
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 03-236
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-10

CONDITIONS: Diphtheria; Hepatitis B; Pertussis; Poliomyelitis; Tetanus
Keywords: umbilical cord blood, vaccine, pregnant women
MeSH Terms: conditions — Diphtheria; Hepatitis B; Whooping Cough; Poliomyelitis; Tetanus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To evaluate and standardize umbilical cord specimen collection and laboratory procedures to evaluate cellular and serological immune responses in neonates and young infants

DETAILED DESCRIPTION:
To evaluate: 1) The procedures for obtaining umbilical cord blood; 2) the methods for ensuring immune cell viability, freezing, and shipping; 3) the conditions for optimization of immune cell isolation procedures.

ELIGIBILITY:
Inclusion Criteria:

For the portion of the pilot study conducted at the UCLA CVR, an umbilical cord blood sample will be obtained from approximately 8 to 12 healthy pregnant women who are delivering neonates at the Obstetrical delivery ward of Harbor- UCLA Medical Center. Informed consent will not be obtained because the blood will be obtained after delivery from a clamped umbilical cord attached to the placenta (afterbirth) that otherwise would be discarded.

Exclusion Criteria:

A cord blood sample will not be collected from women who have requested special arrangements for a cord blood registry service.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Study Completion 2005-02

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Center For Vaccine Research, Torrance, California, United States